CLINICAL TRIAL: NCT05804617
Title: Dome-type (Modified C-incision) Extracorporeal Manual Morcellation During Laparoscopic Uterine Surgery: A Retrospective Analysis
Brief Title: Dome-type (Modified C-incision) Manual Morcellation During Laparoscopic Uterine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202206083RINB
Record Dates: First submitted 2023-02-20; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2022-09

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgeon group (Placebo Comparator): Dome-type morcellation performed by one skillful surgeon
  Interventions: Procedure: Dome-type (Modified C-incision) manual morcellation
- Trainee group (Active Comparator): Dome-type morcellation performed by trainees (residents) under supervision
  Interventions: Procedure: Dome-type (Modified C-incision) manual morcellation

INTERVENTIONS:
Procedure: Dome-type (Modified C-incision) manual morcellation — Morcellation performed by surgeon or trainee

SUMMARY:
In-bag manual morcellation is a safe alternative procedure after FDA's discouragement of electronic power morcellator. The traditional wedging (V-type incision) or semicircular coring (C-type incision or ExCITE) method are the most common morcellation techniques. For beginners, it is somehow not that easy to get familiar with these methods. No teaching or learning experiences were reported. Therefore, we developed a dome-type (modified C-incision) technique to manually morcellate uteri leiomyoma or uterus at the time of laparoscopic surgery and report perioperative outcomes and the learning experiences of our residents for this technique from our two years of experience.

DETAILED DESCRIPTION:
Background: In-bag manual morcellation is a safe alternative procedure after FDA's discouragement of electronic power morcellator. The traditional wedging (V-type incision) or semicircular coring (C-type incision or ExCITE) method are the most common morcellation techniques. For beginners, it is somehow not that easy to get familiar with these methods. No teaching or learning experiences were reported.

Objective: To describe using a dome-type (modified C-incision) technique to manually morcellate uteri leiomyoma or uterus at the time of laparoscopic surgery and report perioperative outcomes and the learning experiences of our residents for this technique from our two years of experience.

Study Design: Retrospective review of consecutive laparoscopic myomectomies or hysterectomies performed between May 2020 and September 2022 in which the specimen was manually morcellated using the dome-type technique by surgeon or trainees.

ELIGIBILITY:
Inclusion Criteria:

* Women at any age undergoing laparoscopic surgeries with dome-type morcellation

Exclusion Criteria:

* Women with extremely huge specimen (>2000 gm)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Morcellation speed | During procedure
  Weight of specimen (gram) divided by morcellation time (minute)

SECONDARY OUTCOMES:
Age | Before procedure
  Age
BMI (kg/m2) | Before procedure
  BMI
Abdominal surgical history | Before procedure
  Any abdominal surgical history, e.g., Cesarean section, myomectomy, appendectomy...
Stiffness | During procedure
  Categorize to soft or hard
Umbilical wound size (cm) | During procedure
  Umbilical wound size
Pathology | 1 week (after the pathologic report being released)
  Final pathologic result, e.g., leiomyoma, adenomyosis...

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Hau Chen, PhD, Principal Investigator — Department of Obstetrics and Gynecology, National Taiwan University Hospital, Taipei, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan